CLINICAL TRIAL: NCT03440723
Title: Inter-examiner Agreement of a Novel Device for the Measurement of Cervical Dilation in Labor: A Randomized Controlled Trial
Brief Title: DilaCheck Cervical Dilation Measurement Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elm Tree Medical Inc. (Industry)
Collaborators: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 16F.270
Record Dates: First submitted 2018-02-07; First posted 2018-02-22 (Actual); Results first posted 2021-06-22 (Actual); Last update posted 2021-06-22 (Actual); Status verified 2021-05

CONDITIONS: Cervical Dilation; Labor Pain; Labor Fast; Labor; Irregular
Keywords: Cervical Dilation; Dilation; Sterile vaginal examination
MeSH Terms: conditions — Labor Pain; Dilatation, Pathologic

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial in which participants are randomly assigned to one of two arms, control or treatment
Masking Description: Masking is not possible since physicians and participants will know whether they are using the device or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Standard Dilation Exam (Active Comparator): Participants receive two standard digital cervical dilation examinations conducted by two different physicians.
  Interventions: Diagnostic Test: Cervical dilation examination
- Dilation Exam with DilaCheck (Experimental): Participants receive two cervical dilation examinations using DilaCheck devices conducted by two different physicians.
  Interventions: Device: DilaCheck

INTERVENTIONS:
Device: DilaCheck — Measuring device for the measurement of cervical dilation
  Arms: Dilation Exam with DilaCheck
Diagnostic Test: Cervical dilation examination — Sterile vaginal examination using subjective methods for measurement of cervical dilation
  Arms: Standard Dilation Exam

SUMMARY:
Trial to compare the interexaminer agreement between two cervical dilation examinations conducted by Labor and Delivery physicians when using standard methods versus DilaCheck device.

DETAILED DESCRIPTION:
The trial seeks to compare the DilaCheck device with standard digital cervical dilation examinations. 50 laboring female participants will be enrolled with 25 randomly assigned to the control arm and 25 to the treatment (DilaCheck) arm. Each participant will receive two cervical dilation examinations from two separate physicians. The main outcome measure is agreement between the two cervical dilation measurements. Secondary outcomes include ease of use of the device and pain levels.

ELIGIBILITY:
Inclusion Criteria:

* The research population is pregnant women in the first stage of labor. Subjects eligible for inclusion in the study must be: pregnant women who are admitted to a Labor and Delivery unit for management or induction of labor in the first stage of labor, are able to give informed consent, are 18 years of age or greater, speak English, and have a gestational age greater than or equal to 37 weeks (i.e. term pregnancy). Patients are only consented if they have adequate pain control, either because they are not yet in labor (i.e. are admitted for an induction of labor) or have a functioning epidural.

Exclusion Criteria:

* Exclusion criteria include progression to the second stage of labor (i.e. known dilation of ten centimeters), known rupture of membranes, any condition that renders labor unsafe for the patient (e.g. cardiac conditions, pulmonary hypertension) and any other condition that necessitates an emergent or urgent cesarean section (e.g. non-reassuring fetal status, placental abruption, hemorrhage, cord prolapse). All participants are necessarily female due to the subject matter. Given the vulnerability of pregnant patients under the age of 18, this study will exclude children. There are no restrictions on eligibility based on race or ethnicity.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2020-01-06 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Martin EL, Firman B, Berghella V. Novel device vs manual examinations for the measurement of cervical dilation in labor: a randomized controlled trial. Am J Obstet Gynecol MFM. 2021 May;3(3):100328. doi: 10.1016/j.ajogmf.2021.100328. Epub 2021 Feb 11. PMID 33582306

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment finalized at 42 due to COVID
Period: Overall Study
Arm/Group | Standard Dilation Exam | Dilation Exam With DilaCheck
Started | 21 | 21
Completed | 21 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard Dilation Exam | Dilation Exam With DilaCheck | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.8 (5.0) | 29.1 (5.6) | 28 (5.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 21 | 42
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 5
  Not Hispanic or Latino | 18 | 19 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 4 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 9 | 24
  White | 6 | 7 | 13
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 21 | 42

OUTCOME MEASURES:

1. Primary Outcome: Interexaminer Agreement
Description: Agreement between 2 cervical dilation measurements taken by 2 different physicians. If the measurements are the same, the outcome is "agree." If the measurements are different, the outcome is "disagree."
Time Frame: Immediate upon examination
Population: All enrollees
Measure: Count of Participants; unit: Participants
Arm/Group | Standard Dilation Exam | Dilation Exam With DilaCheck
Number analyzed (Participants) | 21 | 21
Participants | 9 | 4

2. Secondary Outcome: Pain With Examination
Description: Scores on a Scale. Subjective experience of pain during dilation examinations as measured by scores on a scale given to patient participants following the cervical dilation examinations. The pain measurement is a scale of 1 to 10 with 1 being no pain and 10 being extreme pain. The participant enters a number from 1 to 10 on the survey.
Time Frame: Immediate within 5 minutes of examinations
Population: all enrollees
Measure: Mean (Standard Deviation); unit: score on pain scale
Arm/Group | Standard Dilation Exam | Dilation Exam With DilaCheck
Number analyzed (Participants) | 21 | 21
score on pain scale | 2.8 (2.8) | 3.1 (2.9)

3. Secondary Outcome: Ease of Use
Description: Ease of Use of the device as reported by physician users on a paper survey administered to them. Reported is number of physicians who reported device is easy to use.
Time Frame: Upon conclusion of the trial, <3 months from time of last examination with device
Population: All providers who participated in the trial completed the survey
Measure: Count of Participants; unit: Participants
Groups:
- Providers Participating in Trial: 10 providers participated in the trial providing examinations and provided feedback on ease of use of the device.
Arm/Group | Providers Participating in Trial
Number analyzed (Participants) | 10
Participants | 7

ADVERSE EVENTS:
Time Frame: 30-90 minutes
Arm/Group | Standard Dilation Exam | Dilation Exam With DilaCheck
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 0/21 | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-01): https://cdn.clinicaltrials.gov/large-docs/23/NCT03440723/Prot_SAP_000.pdf